CLINICAL TRIAL: NCT07201701
Title: Is CYP24A1 Heterozygosity a Risk Factor for Nephrolithiasis?
Acronym: HETEROCYP
Status: Not yet recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL25_0507; 2025-A01749-40 (Other: ID-RCB)
Record Dates: First submitted 2025-09-22; First posted 2025-10-01 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Nephrolithiasis
Keywords: CYP24A1 heterozygous; Nephrolithiasis; CYP24A1 homozygous, and compound heterozygous; Nephrocalcinosis
MeSH Terms: conditions — Nephrolithiasis; Nephrocalcinosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients carriers of a heterozygous CYP2A1 mutation: Patients carriers of a heterozygous CYP2A1 mutation with or without symptoms: history of nephrocalcinosis or nephrolithiasis
  Interventions: Biological: Supplementary blood samples for PBMC analysis at V2
- Patients carriers of homozygous, and compound heterozygous CYP2A1 mutation: Patients carriers of homozygous, and compound heterozygous CYP2A1 mutation with or without symptoms: history of nephrocalcinosis or nephrolithiasis
  Interventions: Biological: Supplementary blood samples for PBMC analysis at V2

INTERVENTIONS:
Biological: Supplementary blood samples for PBMC analysis at V2 — Supplementary blood (serum and plasma) and urines samples for bio collection at V3

SUMMARY:
Biallelic loss-of-function variants in CYP24A1 have been identified as a common genetic cause of autosomal recessive hypercalcemia (ARH, ORPHA 300547, 1 in 80,000 live births), characterized by low PTH (parathyroid hormone) levels, a high 25-OH D/24,25-(OH)₂D ratio, and susceptibility to vitamin D intoxication.

In humans, heterozygous pathogenic variants in CYP24A1 have been proposed both as responsible for an autosomal dominant disorder and as a risk factor for nephrolithiasis, but the rarity and heterogeneity of human data prevent a definitive answer to this crucial question.

Nephrolithiasis is a complex disease in which nutritional factors - particularly sodium and protein intake (leading to hypercalciuria) - play a key role. It also has a heritability of 50%, suggesting the involvement of many genetic susceptibility factors, as well as monogenic forms (mainly autosomal recessive, but also dominant or X-linked), which have been identified in 10-20% of patients.

The increasing prevalence of nephrolithiasis, affecting approximately 10% of the general population over a lifetime, has a significant financial impact on healthcare systems and imposes a major burden of morbidity, justifying further investigation into the genetic underpinnings of nephrolithiasis.

The goal of the HeteroCYP project is to improve understanding of the phenotypes associated with heterozygous, compound heterozygous, and homozygous variants of CYP24A1 by comparing clinical and biological outcomes in patients according to their mutation type

ELIGIBILITY:
Inclusion Criteria:

Group 1: Heterozygous Patients

* Aged between 2 and 90 years
* Weight > 12 kg
* Carriers of a heterozygous CYP24A1 mutation
* With or without symptoms: history of nephrocalcinosis or kidney stones

Group 2: Homozygous / Compound Heterozygous Patients

* Aged between 2 and 90 years
* Weight > 12 kg
* Carriers of a homozygous or compound heterozygous CYP24A1 mutation
* With or without symptoms: history of nephrocalcinosis or kidney stones

Exclusion Criteria:

* Individuals unable to collect 24-hour urine
* Individuals unable to be available for a full day in a day hospital (HDJ)
* Pregnant, postpartum, or breastfeeding women
* Individuals deprived of liberty by judicial or administrative decision
* Individuals receiving psychiatric care
* Individuals admitted to a healthcare or social institution for reasons other than participation in research
* Adults under legal protection (guardianship or trusteeship)
* Individuals not affiliated with a social security system or not benefiting from an equivalent scheme

Ages: 2 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study focuses on patients who are CYP24A1 heterozygous, CYP24A1 homozygous, or compound heterozygous.
Sampling Method: Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of nephrolithiasis in patients who are CYP24A1 heterozygous and homozygous (or compound heterozygous) | Visit 2 (at least 24 hours after baseline)
  Prevalence of nephrolithiasis (based on imaging) in patients who are CYP24A1

CONTACTS AND LOCATIONS:
Overall Officials: Justine Pr BACCHETTA, Principal Investigator — Hospices Civils de Lyon
Locations (2):
- France (2):
  - Hôpital Femme Mère Enfant, Bron
  - Hôpital Edouard Herriot, Lyon